CLINICAL TRIAL: NCT07195097
Title: A Prospective Study to Evaluate the Efficacy of Silodosin 8 mg as an on-Demand, Reversible, Nonhormonal Oral Contraceptive for Males:
Brief Title: Sildosin as a Male Contraceptive Non Hormonal
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohamed Farag Ali, Lecturer and consultant of urology, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC 5-10-2024
Record Dates: First submitted 2025-07-14; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Contraception Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sildosin arm (Active Comparator): Oral intake of sildosin
  Interventions: Drug: Oral intake of sildosin
- Placebo arm (Placebo Comparator): Oral intake of placebo
  Interventions: Other: Oral intake of placebo

INTERVENTIONS:
Drug: Oral intake of sildosin — Oral intake of sildosin in male non hormonal contraception
  Arms: Sildosin arm
Other: Oral intake of placebo — Intake of placebo to compare effecacy of other group
  Arms: Placebo arm

SUMMARY:
In all, 200 healthy, sexually active, fertile male candidates will be assigned 100 in silodosin group and 100 in placebo group. Males using other contraceptive methods will be excluded. Follow up data of total spermatozoa per ejaculate, semen volume and Post-ejaculation urinalysis after 2, 6 and 12 weeks of the studied groups will be recorded. The various side effects reported in the study groups after 12 weeks from the start of the study will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* male sexually active

Exclusion Criteria:

* male on oral contraceptives Male with female partner on contraceptives

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 200 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate in people treated with sildosin as a male contraceptive | 3 months
  Pregnancy rate in people treated with sildosin as a male contraceptive treatment